CLINICAL TRIAL: NCT02060123
Title: A Randomized, Wait-list Controlled Trial of a Qigong Intervention Program on Telomerase Activity and Psychological Stress in Abused Chinese Women
Brief Title: Qigong Intervention Program for Abused Chinese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Agnes Tiwari, Professor and Head, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UW 12-555
Record Dates: First submitted 2014-02-06; First posted 2014-02-11 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Abused Women
Keywords: Qigong; Telomerase; Perceived stress; RCT; Chinese; Abused women; intervention; Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Qigong training (Experimental): a total of 103 hours over a period of 5.5 months, consisting of:
  * Group learning and practice: a 2-hour qigong exercise training session will be provided by a qigong master twice a week for six consecutive weeks (24 hours),
  * Weekly group follow-up: a 1-hour qigong exercise will be conducted with reinforcement of learning and remedial teaching by a qigong master once a week for four consecutive months (16 hours) after the group learning and practice, and
  * Self-practice: participant will engage in qigong exercise for 30 minutes every day for the whole intervention period lasting 5.5 months (63 hours).
  Interventions: Behavioral: Qigong training
- Wait-list control- Health talks (Other): Monthly health education talks unrelated to qigong will be provided starting from the point when the intervention group starts the qigong weekly follow-up.Once the intervention group has completed the qigong intervention program, the wait-list control group will receive the qigong exercise training.
  Interventions: Other: Wait-list control- Health talks

INTERVENTIONS:
Behavioral: Qigong training — a total of 103 hours over a period of 5.5 months, consisting of:
  * Group learning and practice: a 2-hour qigong exercise training session will be provided by a qigong master twice a week for six consecutive weeks (24 hours),
  * Weekly group follow-up: a 1-hour qigong exercise will be conducted with reinforcement of learning and remedial teaching by a qigong master once a week for four consecutive months (16 hours) after the group learning and practice, and
  * Self-practice: participant will engage in qigong exercise for 30 minutes every day for the whole intervention period lasting 5.5 months (63 hours).
  Arms: Qigong training
Other: Wait-list control- Health talks — Monthly health education talks unrelated to qigong will be provided starting from the point when the intervention group starts the qigong weekly follow-up.Once the intervention group has completed the qigong intervention program, the wait-list control group will receive the qigong exercise training.
  Arms: Wait-list control- Health talks

SUMMARY:
The purpose of this study is to evaluate the effect of a qigong intervention program on telomerase activity in Chinese women with a history of intimate partner violence.

DETAILED DESCRIPTION:
Qigong is a mind-body exercise rooted in the paradigm of traditional Chinese medicine, aiming to achieve a harmonious flow of energy (qi) in the body through gentle movements and is thus considered as a holistic health practice towards promoting physical and mental well-being and improving longevity. It was suggested that qigong exercise, as a stress management strategy, could be effective in improving psychological symptoms, as well as enhancing cellular telomerase activity by reducing oxidative stress level and regulating immune response.

The study is to evaluate the effects of a qigong intervention on telomerase activity and pro-inflammation cytokines, perceived stress, perceived coping, and depressive symptoms in Chinese women with a history of intimate partner violence. The study design is a randomized, wait-list controlled design with intervention and wait-list control groups. A total of 240 Chinese abused women will be recruited. The qigong intervention program consists of: (i) a 2-hr group qigong training twice a week for 6 weeks; (ii) weekly group follow-up of a 1-hour group qigong exercise for 4 months; and (iii) self-practice of qigong exercise for 30 minutes each day throughout the intervention period lasting 5.5 months. It is hypothesized that the participants in the intervention group will have higher levels of telomerase activity and perceived coping, and lower levels of pro-inflammation cytokines, perceived stress, and depressive symptoms, on completion of a qigong intervention program, compared to abused Chinese women in the wait-list control group.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* willing to undertake the qigong intervention program,
* available for all testing points,
* receptive to random allocation, and
* assessed to be abused by an intimate partner in the preceding year or longer, based on the Chinese Abuse Assessment Screen.

Exclusion Criteria:

* had participated in qigong training or other mind body intervention within the previous 6 months, or
* have serious medical conditions that might limit their participation in qigong exercise (based on our previous experience, such conditions include cancer, severe obesity, narcolepsy, major depressive disorder, schizophrenia), or
* have psychiatric disorders, or
* use medication or other psychological intervention for stress, or
* are abused by someone who is not their intimate partner.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2014-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in telomerase activity | pre-intervention (baseline) and post-intervention (5.5 months later)
  For each participant, 10 ml of peripheral blood will be collected for measurements of telomerase activity at two time points: pre-intervention (T0) and post-intervention (T2) in the intervention group, as well as in wait-list control group before qigong training.

SECONDARY OUTCOMES:
Change in level of pro-inflammatory cytokines | pre-intervention (baseline) and post-intervention (5.5 months later)
  The peripheral blood plasma will also be analyzed for pro-inflammation cytokines TNF-alpha and IL-6 levels.
Change in perceived stress | pre-intervention (baseline), post-training (6 weeks later) and post-intervention (5.5 months later)
  The 10-item Perceived Stress Scale (PSS), the most widely used psychological instrument for measuring the perception of stress, will be used to assess the degree to which situations in life are perceived by the participant as stressful during the past month.
Change in perceived coping | pre-intervention (baseline), post-training (6 weeks later) and post-intervention (5.5 months later)
  The Perceived Coping Scale (PCS) will be used to assess the types and perceived effectiveness of each of the 13 specific strategies used by the participant in dealing with violence perpetrated by her intimate partner.
Change in depressive symptoms | pre-intervention (baseline), post-training (6 weeks later) and post-intervention (5.5 months later)
  The Chinese version of the Beck Depression Inventory version II (BDI-II) will be used to assess depressive symptoms in the previous two weeks.
Change in sleep disturbance | pre-intervention (baseline), post-training (6 weeks later) and post-intervention (5.5 months later)
  The Chinese version of the General Sleep Disturbance Scale (GSDS), a 21-item questionnaire, will be used to measure participants' sleep disturbance.

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Tiwari, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- HKSKH Lady MacLehose Center, Hong Kong, China

REFERENCES:
- [Background] Ho RT, Chan JS, Wang CW, Lau BW, So KF, Yuen LP, Sham JS, Chan CL. A randomized controlled trial of qigong exercise on fatigue symptoms, functioning, and telomerase activity in persons with chronic fatigue or chronic fatigue syndrome. Ann Behav Med. 2012 Oct;44(2):160-70. doi: 10.1007/s12160-012-9381-6. PMID 22736201
- [Background] Zhang GD. The impacts of 48-form tai chi chuan and yi qi yang fei gong on the serum levels of IgG, IgM, IgA, and IgE in human. Journal of Beijing Institute of Physical Education. 1990;4:12-4.
- [Background] Jahnke R, Larkey L, Rogers C, Etnier J, Lin F. A comprehensive review of health benefits of qigong and tai chi. Am J Health Promot. 2010 Jul-Aug;24(6):e1-e25. doi: 10.4278/ajhp.081013-LIT-248. PMID 20594090
- [Derived] Cheung DST, Chau PH, Yeung WF, Deng W, Hong AWL, Tiwari AFY. Assessing the effect of a mind-body exercise, qigong Baduanjin, on sleep disturbance among women experiencing intimate partner violence and possible mediating factors: a randomized-controlled trial. J Clin Sleep Med. 2021 May 1;17(5):993-1003. doi: 10.5664/jcsm.9102. PMID 33551021
- [Derived] Hameed M, O'Doherty L, Gilchrist G, Tirado-Munoz J, Taft A, Chondros P, Feder G, Tan M, Hegarty K. Psychological therapies for women who experience intimate partner violence. Cochrane Database Syst Rev. 2020 Jul 1;7(7):CD013017. doi: 10.1002/14651858.CD013017.pub2. PMID 32608505
- [Derived] Cheung DST, Deng W, Tsao SW, Ho RTH, Chan CLW, Fong DYT, Chau PH, Hong AWL, Fung HYKY, Ma JLC, Tiwari AFY. Effect of a Qigong Intervention on Telomerase Activity and Mental Health in Chinese Women Survivors of Intimate Partner Violence: A Randomized Clinical Trial. JAMA Netw Open. 2019 Jan 4;2(1):e186967. doi: 10.1001/jamanetworkopen.2018.6967. PMID 30646209
- [Derived] Tiwari A, Chan CL, Ho RT, Tsao GS, Deng W, Hong AW, Fong DY, Fung HY, Pang EP, Cheung DS, Ma JL. Effect of a qigong intervention program on telomerase activity and psychological stress in abused Chinese women: a randomized, wait-list controlled trial. BMC Complement Altern Med. 2014 Aug 15;14:300. doi: 10.1186/1472-6882-14-300. PMID 25127878